CLINICAL TRIAL: NCT05129046
Title: Neutrophil-to-Lymphocite Ratio (NLR) and C-reactive Protein (CRP) as New Markers in Diagnosis and Prediction of Surgical and Oncological Outcomes in Colorectal Cancer
Brief Title: Neutrophil-to-Lymphocite Ratio (NLR) and C-reactive Protein (CRP) as New Markers in Diagnosis and Prediction of Colorectal Cancer
Acronym: NelyCre
Status: Recruiting | Type: Observational
Sponsor: Azienda Ospedaliera SS. Antonio e Biagio e Cesare Arrigo di Alessandria (Other)
Responsible Party: Principal Investigator, Igor Monsellato, Principal Investigator, Azienda Ospedaliera SS. Antonio e Biagio e Cesare Arrigo di Alessandria
Other Study IDs: ASO.ChirGen.21.03
Record Dates: First submitted 2021-11-09; First posted 2021-11-22 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; robotic surgery; cancer biomarkers; interleukines; NLR; CRP
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Colorectal cancer (CRC) is the second leading cause of cancer-related death in the Western world. Overall survival (OS) remains poor, with 50% estimated 5-year survival. In Italy, current estimates indicate that in 2020 a number of 43.700 patients have been affected by colorectal cancer, with an increasing of diagnosed cases in both men and women. It is clear that it is worthwhile to investigate the evaluation of colorectal cancer which could reflect a different spread of screening programs or be the effect of different timing in the start of the programs themselves. To improve the overall survival of colorectal cancer patients, robust biomarkers for screening and predicting disease recurrence could help identify high-risk patients, facilitate a close patient follow-up, and decide appropriate treatment regimens during the postoperative care. Colonoscopy remains the most efficient method for detecting CRC, yet its general application in the setting of screening is limited due to the uncomfortable experience and the high costs. accumulating studies have revealed the potential of systemic inflammatory markers such as C-reactive protein (CRP), albumin, neutrophils, platelets, and lymphocytes, and also biomarker combination ratios [(eg, CRP-albumin ratio (CAR), neutrophil-lymphocyte ratio (NLR), and platelet-lymphocyte ratio (PLR)] as prognostic biomarkers in different cancers, including CRC. Chronic inflammation affects all stages of tumor development. Several studies have shown that various preoperative markers reflecting systemic inflammatory response, including NLR and CRP ratio, offer predictive potential for postoperative morbidity and mortality in CRC patients. However, several issues require addressing prior to the adoption of these inflammatory markers in the clinical practice for CRC patients undergoing surgery: a) the combination of inflammatory factors that might be best in predicting oncological outcomes in colorectal cancer patients remains unclear; b) previous studies for systemic inflammatory markers have mainly interrogated their prognostic potential for oncological outcomes but have not laid emphasis for evaluating their predictive value for postoperative complications; c) there is a lack of consensus on the cut-off thresholds used for each marker for determining mortality risk resulting from surgical and oncological outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Histologically-proven adenocarcinoma of the colon or the rectum
* Eligible for a resective surgery by minimally-invasive (standard or robotic-assisted laparoscopic procedure, all robotic systems will be accepted) or open approach
* Able to give written informed consent

Exclusion Criteria:

* Squamous carcinoma of the anal canal
* History of psychiatric or addictive disorder or other medical condition that, in the opinion of the investigator, would preclude the patient from meeting the trial requirements
* Pregnancy
* Unable to give free informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from colorectal cancer will be identified after endoscopy and screened for inclusion into the study once referred to the colorectal surgeon. Patients will be approached for possible recruitment following diagnosis and radiological staging, provided they fulfil the inclusion/exclusion criteria. Patients will be provided with verbal and written details. A verbal explanation of the trial will be provided by a medically qualified member of the healthcare team for the patient to consider.
  Patients who accept to participate in, will then be formally assessed for eligibility and invited to provide informed, written consent for their participation in the trial.
  A total of 100 patients will be enrolled in the trial.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
DFS | 5 years
  Disease Free Survival

SECONDARY OUTCOMES:
OS | 5 years
  Overall Survival
Surgical Outcomes | 90 days
  Correlation of changes in NLR, PLR and CAR and ILs following complete surgical resection with postoperative complications

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - SS. Antonio e Biagio e Cesare Arrigo, Alessandria
  - San Raffaele Hospital, Milan